CLINICAL TRIAL: NCT01777516
Title: In Vitro Study to Evaluate the Pharmacodynamic Interaction Between Ticagrelor and Its Active Metabolite (AR-C124910XX) and Their Effects on the Pharmacodynamics of Salicylic Acid : Concentration-antiplatelet Effect Relationships
Brief Title: In Vitro Interaction Between Ticagrelor and Its Active Metabolite and Their Effects on Salicylic Acid
Acronym: In_vitro_PAT
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Korea National Enterprise for Clinical Trials (Other)
Responsible Party: Principal Investigator, Hyeong-Seok Lim, Associate Professor of the Department of Pharmacology and Therapeutics, Asan Medical Center
Other Study IDs: AsanMC_CPT_PAT_2012; A070001 (Other Grant/Funding Number: Korea National Enterprise For Clinical Trials)
Record Dates: First submitted 2013-01-22; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Diseases
Keywords: Platelet Aggregation; Cardiovascular Diseases; Salicylic Acid
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Plasma and white blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers: 1 group with no treatment : They provide the blank plasma to be used at in vitro study.

SUMMARY:
This is a in-vitro study to evaluate the pharmacodynamic interaction between ticagrelor and its active metabolite (AR-C124910XX) and their effects on the pharmacodynamics of salicylic acid. The study consist of two parts of in-vitro study as follows;

* Part 1 : in-vitro study to evaluate the pharmacodynamic interaction between ticagrelor and its active metabolite.
* Part 2 : in vitro study to evaluate the pharmacodynamic interaction between ticagrelor and its active metabolite and their effect on the pharmacodynamics of salicylic acid on platelet aggregation tests with the agonist of arachidonic acid.

DETAILED DESCRIPTION:
This is a in-vitro study to evaluate the pharmacodynamic interaction between ticagrelor and its active metabolite (AR-C124910XX) and their effects on the pharmacodynamics of salicylic acid. The study consist of two parts of in-vitro study as follows;

* Part 1 : in-vitro study to evaluate the pharmacodynamic interaction between ticagrelor and its active metabolite. Platelet aggregation tests with the agonist of adenosine diphosphate(ADP) will be assessed on the in-vitro mixtures of blank plasma and randomized paired concentrations of ticagrelor + AR-C124910XX.
* Part 2 : in vitro study to evaluate the pharmacodynamic interaction between ticagrelor and its active metabolite. Platelet aggregation tests with the agonist of arachidonic acid will be assessed on the in-vitro mixtures of blank plasma plus randomized paired concentrations of ticagrelor and AR-C124910XX and the invitro mixtures with blank plasma and ticagrelor + AR-C124910XX + salicylic acid.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with body weight more than 50 kg and within 20% of the ideal body weight: ideal body weight = (height[cm] - 100)*0.9.
* Subjects who have received and understood completely the information regarding the current study and given written informed consents to voluntarily participate in the study and followed all instructions specified in the protocol.

Exclusion Criteria:

* Subjects who have a history or presence of any clinically significant diseases.
* Subjects who have any congenital or acquired haematological diseases.
* Subjects who had whole blood donation within the last 2 months and component blood donation within the last month.
* Subject who took any concomitant medication including non-steroidal antiinflammatory drugs(NASIDs) and vitamins currently or within 7 days prior to blood sampling.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation(%) of the in vitro mixtures of blank plasma and drugs of the randomized paired concentrations | The tolerability of volunteers after blood sampling will be followed for the duration of hospital stay, an expected average of 5 hours.
  Plasma which were collected from healthy volunteers were used to make mixtures of drugs, ticagrelor, AR-C124910XX and salicylic acid. ADP and arachidonic acid were used as the agonists of platelet aggregation.

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, M.D., PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea